CLINICAL TRIAL: NCT02292992
Title: The Difference of Lung Volume Change Detected by Electrical Impedance Tomography (EIT) Between Noninvasive Positive-pressure Ventilation (NIPPV) Support by Nasal Pillow and High Flow Nasal Cannula in Post-extubation Patients
Brief Title: Lung Volume Change Between Noninvasive Positive Pressure Ventilation by Nasal Pillow and High Flow Nasal Cannula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14MMHIS167
Record Dates: First submitted 2014-10-27; First posted 2014-11-18 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Failure
Keywords: Electrical impedance tomography; Nasal Pillow Continuous Positive Airway Pressure(CPAP); High Flow Nasal Cannula; extubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nasal pillow CPAP (Experimental): Nasal pillow CPAP
  Interventions: Device: Nasal Pillow CPAP

INTERVENTIONS:
Device: Nasal Pillow CPAP — Nasal Pillow CPAP in extubated patients

SUMMARY:
The difference of lung volume change will be monitored by electrical impedance tomography before and after use of noninvasive positive pressure ventilation by nasal pillow and high flow nasal cannula in post-extubation patients.

DETAILED DESCRIPTION:
Electrical impedance tomography can effectively monitor the lung volume change in ICU patients who were under mechanical ventilator or noninvasive positive pressure ventilator support. Continuous positive airway pressure (CPAP) support by nasal pillow and high flow nasal cannula can improve inspiratory function in extubated patients . However, the extent of lung volume change or functional residual volume (FRC) change by using these two devices were never surveyed before in extubated patients. The investigators will check end-expiratory lung volume (EELV) ,anterior, medio-anterior, medio-posterior and posterior EELV by electrical impedance tomography after use of these two devices in extubated patients.

ELIGIBILITY:
Inclusion Criteria:

* >20 y/o
* Any extubated patients after tolerating spontaneous breathing trial

Exclusion Criteria:

* Presence of tracheostomy
* Recent facial trauma
* Active gastro-intestinal bleeding
* Do-not-intubate status and
* Planned use of BiPAP after extubation.
* Patients with unstable spinal lesions or fractures.
* BMI> 50
* Patients with a cardiac pacemaker
* Burn injury with skin defect

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
• End-expiratory lung volume (EELV) determined by electrical impedance tomography after high flow nasal cannula and nasal pillow CPAP | at day 1

SECONDARY OUTCOMES:
Anterior, medio-anterior, medio-posterior and posterior EELV at each time | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Lee Chao-Hsien, MD, Principal Investigator — +886975835770 l49428@mmh.org.tw
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan